CLINICAL TRIAL: NCT04721210
Title: A Prospective Randomized, Blind, Placebo-controlled Trial "The Effectiveness of Transcranial Magnetic Stimulation of Supplementary Motor Area (SMA) in Patients With Bladder Hypersensitivity and Bladder Pain
Brief Title: The Effectiveness of Transcranial Magnetic Stimulation of Supplementary Motor Area (SMA) in Patients With Bladder Hypersensitivity and Bladder Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Joint-Stock Company North-West Center for Evidence-Based Medicine, Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1/2021
Record Dates: First submitted 2021-01-13; First posted 2021-01-22 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Bladder Hypersensitivity
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Frequency of 1 Hz (Experimental): continuous stimulation with a frequency of 1 Hz, 2000 pulses, 10 days-daily;
  Interventions: Other: Transcranial magnetic stimulation
- Frequency of 10 Hz (Experimental): continuous stimulation with a frequency of 10 Hz-10 seconds with a pause of 50 seconds, 2000 pulses, 10 days-daily;
  Interventions: Other: Transcranial magnetic stimulation
- Continuous stimulation placebo (Placebo Comparator): continuous stimulation placebo
  Interventions: Other: Transcranial magnetic stimulation

INTERVENTIONS:
Other: Transcranial magnetic stimulation — The investigated method is called transcranial magnetic The impact on the SMA will be made using a special inductor of the "double conical coil" type. Navigation will be carried out through the use of the international system "10-20%". The threshold of motor response will be determined by stimulating the motor area of the legs with the intensity of stimulation necessary to trigger a motor response with an amplitude of more than 50 mv.

SUMMARY:
The main hypothesis of this study is that transcranial magnetic neuromodulation can correct the symptoms of hypersensitivity and bladder pain. The investigators assume that under the influence of transcranial magnetic stimulation, both the subjective state of patients assessed by standardized questionnaires and the objective parameters assessed by invasive and non-invasive urodynamic studies will be improved. In this study, two protocols for magnetic stimulation of the supplementary motor area (SMA) will be compared with each other and with placebo. The investigators expect to determine the dependence of the therapeutic effect on the applied stimulation protocol.

DETAILED DESCRIPTION:
The aim of the study is to test the hypothesis that the use of the magnetic stimulation method SMA in patients with symptoms of bladder hypersensitivity and bladder pain will help to reduce the clinical and urodynamic signs of these pathological conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years;
2. Signed informed consent;
3. The presence of OAB symptoms: urinary frequency, nocturia, urgency and urge incontinence; discomfort during filling the bladder, pain in the projection of the bladder over the womb.
4. Resistance to standard therapy for bladder hypersensitivity and bladder pain.

Exclusion Criteria:

1. The patient, who have been implanted devices that control physiological functions (a pacemaker, a device for deep brain stimulation and chronic epidural brain stimulation, a cochlear implant).
2. Convulsive attacks in the anamnesis;
3. Taking medications that may trigger the risk of seizures;
4. Pregnancy or suspicion on it;
5. The presence in the patient's body of metal elements or objects made with the use of ferromagnets (joint prostheses, eye prostheses, tattoos made using metal ink, surgical clips, staples and other metal suture materials, etc.)
6. Chronic cardiovascular and cerebrovascular diseases in the stage of decompensation or recent acute conditions (myocardial infarction, brain stroke, etc.)
7. A history of injuries associated with impaired conduction along the pathways of the brain and spinal cord;
8. The presence of detrusor hyperactivity patterns according to the preliminary multichannel urodynamic study;
9. The presence of infravesical obstruction in men, determined by uroflowmetry (obstructive urination curve according to the Liverpool nomogram);
10. The postvoid residual volume (more than 100 ml);
11. The presence of urinary tract infection;
12. A history of cancer;

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-01-20 (Estimated); Study Completion 2022-01-20 (Estimated)

PRIMARY OUTCOMES:
VAPS change score | Baseline, 4, 12, 24, 48 weeks
  VAPS is a continuous scale in the form of a horizontal or 10 cm (100 mm) long and located on it with two extreme points "no pain" and "the strongest pain that can be imagined
OAB-Q SF change score | Baseline, 4, 12, 24, 48 weeks
  Individual participant change score on the Overactive Bladder Questionnaire short-form (OAB-q SF) will be compared between the two cohorts by student's t-test. The OAB-q SF is utilized to assess the impact of OAB symptoms on the patient's life, and has been shown to be responsive to reductions in urinary urgency, frequency and incontinence during transvertebral magnetic neuromodulation therapy. The OAB-q SF questionnaire consists of 19 items divided into a 6-item symptom severity (SS) scale and a 13-item health-related quality of life (HRQL) scale, with both scales ranging from 0 to 100. For the OAB-q SS scale a higher score indicates worse symptom severity while for the OAB-q HRQL scale a higher score indicates better quality of life.
Hospital Anxiety and Depression Scale change score | Baseline, 4, 12, 24, 48 weeks
  The Hospital Anxiety and Depression Scale (HADS) consists of 14 questions: 7 questions assessing anxiety and 7 questions assessing the presence of depression.
Change baseline of micturition episodes per day | Baseline, 4, 12, 24, 48 weeks
  Patients should document how many times they go to the restroom during the day and at night, as well as the loss of urine in stressful situations (coughing, sneezing, laughter, squatting, weightlifting, walking, running), changing liner or absorbent and episodes of urgency and urgency-incontinence. The journal shall be held for a consecutive period of 24 hours, for a minimum of three consecutive days.

SECONDARY OUTCOMES:
Improvement of urodynamic parameters | Baseline, 4, 12, 24, 48 weeks
  Secondary endpoints were evaluated using invasive and non-invasive urodynamic studies: uroflowmetry, filling cystometry, and pressure/flow studies. Invasive urodynamic studies will be performed using a transurethral catheter with 3 lumen transurethral catheter in the bladder and a balloon catheter installed in the vagina or rectum to measure abdominal pressure. The rate of filling the bladder is 30 ml/min in the patient's sitting position on the uroflowmetric chair.

CONTACTS AND LOCATIONS:
Locations (1):
- Joint-Stock Company "North-Western Centre of Evidence-Based Medicine", Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No